CLINICAL TRIAL: NCT06821529
Title: Stereotactic Intracerebral Injection of Autologous Induced Pluripotent Stem Cell-derived Dopamine Progenitor Cells in Patients with Parkinson's Disease
Brief Title: Stereotactic Intracerebral Injection of IPSC-DAPs in Patients with Parkinson's Disease
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: iCamuno Biotherapeutics Ltd. (Industry)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: (2025)LSYD(0172)H
Record Dates: First submitted 2025-02-04; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ICA07 therapy (Experimental): Stereotactic Intracerebral Injection of 4 million iPSC-DAPs into the putamen on each side of the brain .
  Interventions: Biological: ICA07 therapy

INTERVENTIONS:
Biological: ICA07 therapy — 4 million iPSC-DAPs will be administrated into the putamen on each side of the brain

SUMMARY:
Parkinson's disease is a progressive neurodegenerative disorder characterized by high morbidity due to the limited regenerative capacity of dopaminergic neurons in the brain. Current drug treatments primarily manage symptoms but do not halt or reverse neuronal loss. Cellular replacement therapy has emerged as a potential strategy to restore dopaminergic function and address the underlying neuronal deficits. This study aims to evaluate the safety, feasibility, and efficacy of transplanting dopaminergic neurons into the brain to improve motor function and quality of life in patients with advanced Parkinson's disease.

DETAILED DESCRIPTION:
Patients with Parkinson's disease will be treated with autologous induced pluripotent stem cell-derived dopamine progenitor cells (iPSC-DAPs). These cells will be transplanted directly into the striatum to restore dopamine-producing capacity. Patients will be evaluated at 1, 3, 6, 9 and 12 months after transplantation for safety, feasibility, and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Able to sign informed consent and comply with the study protocol
* 39-75 years of age, at the time of signing informed consent
* Diagnosed to be Parkinson's disease patients over 5 years
* Taking levodopa, but with complications of therapy such as wearing off and/or dyskinesia
* At least 3 hours accumulative "off" time per day
* Hoehn and Yahr Stage 2.5 - 4 in the off state at screening
* Dopamine drug responsiveness demonstrated by a positive "on/off" test with at least a 30% improvement on UPDRS III (motor) scale

Exclusion Criteria:

* Patients with the following concomitant conditions or disorders: Epilepsy；Multiple sclerosis；Unable to give consent due to dementia；Atypical Parkinsonism；Genetic Parkinson's disease；Suicidal ideation associated with intent or plan in the past 12 months；History of psychosis；History of subarachnoid hemorrhage；History of stroke or transient ischemic attack
* Patient with unstable vital sign at screening and/or prior to the surgery:
* Estimated Glomerular Filtration Rate (eGFR) < 60 ml/min/1.73m2
* Liver dysfunction, as evidenced by enzymes (AST and ALT) greater than three times the ULN.
* Hematologic abnormality: hemoglobin <10 mg/dL or platelet count < 100,000/mL
* International normalized ratio (INR) ≥ 1.3 not due to a reversible cause
* Patients with autoimmune disorders
* Patients with HIV and/or active HBV or HCV
* Patients who are unable to undergo MRI and PET/CT
* Patients with an expected life expectancy of <1 year
* Patients who have had active malignancies
* Patients currently receive levodopa-carbidopa intestinal gel or apomorphine treatment
* Patients who have history of pallidotomy or thalamotomy or deep brain stimulation (DBS) surgery
* Received cell or gene therapy (autologous or allogeneic) within the previous 12 months
* Participation in an investigational therapeutic or device trial within 30 days of consent
* Women who are pregnant or breast-feeding
* Other conditions that researchers consider not suitable to participate in this study

Ages: 39 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and servility of Treatment-Emergent Adverse Events | From baseline to 12 months post surgery
  Incidence of adverse event (AE), serious adverse event(SAE) is defined as the composite of number and severity of adverse events, regardless of causality, clinical laboratory abnormalities, clinical meaningful changes from baseline

SECONDARY OUTCOMES:
changes in motor function | From baseline to 12 months post surgery
  Changes in motor function that measured by Movement and Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III. TheMDA- UPDRS Part III score ranges from 0 to 132, with higher score indicating greater disability
Changes in the Hoehn and Yahr scale | From baseline to 12 months post surgery
  Hoehn and Yahr scale is used to provide a general estimate of clinical function of PD patients, combining functional deficits (disability) and objective signs (impairment). The Hoehn and Yahr score ranges from 0 to 5, with higher score indicating higher dysfunction of PD patients
Changes in quality of life (QoL) | From baseline to 12 months post surgery
  Measured by Parkinson's Disease Quality of Life Rating Scale (PDQ-39) from baseline to 12 months post surgery.
  PDQ-39 score ranges from 0 to 156 and provides the evidence of the quality of life of a PD patient. The higher the score, the lower the quality of life of PD patients.
Change in PD medication usage | From baseline to 12 months post surgery
  Change in the Parkinson's disease medication usage as defined by the levodopa equivalent daily dose (LEDD)
18-F DAT PET uptake | Baseline, 6 and 12 months post surgery
  Changes in putamen 18F DAT PET uptake that measured by PET/CT

CONTACTS AND LOCATIONS:
Overall Officials: Baorong Zhang, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Gao Chen, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No